CLINICAL TRIAL: NCT04612855
Title: Post-traumatic Neuropathy of the Trigeminal Nerve
Status: Completed | Type: Observational
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Frederic Van der Cruyssen, Prinicipal investigator, KU Leuven
Other Study IDs: S62333
Record Dates: First submitted 2020-10-28; First posted 2020-11-03 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Nerve Injury; Orofacial Pain; Trigeminal Nerve Injuries; Trigeminal Neuropathy
Keywords: post-traumatic trigeminal neuropathic pain
MeSH Terms: conditions — Facial Pain; Trigeminal Nerve Injuries; Trigeminal Nerve Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Painful post-traumatic trigeminal nerve injuries: Patients presenting with painful post-traumatic trigeminal nerve injuries according to the recent ICOP criteria.
  Interventions: Other: Groupwise comparison of primary and secondary outcomes
- Non-painful post-traumatic trigeminal nerve injuries: Patients presenting with non-painful post-traumatic trigeminal nerve injuries according to the recent ICOP criteria.
  Interventions: Other: Groupwise comparison of primary and secondary outcomes
- Temporary nerve injuries: Patients with a trigeminal nerve injury with symptom resolution within 3 months after data of trauma.
  Interventions: Other: Groupwise comparison of primary and secondary outcomes
- Persistent nerve injuries: Patients with a trigeminal nerve injury and complaints persisting longer than 3 months after the trauma.
  Interventions: Other: Groupwise comparison of primary and secondary outcomes

INTERVENTIONS:
Other: Groupwise comparison of primary and secondary outcomes — Statistical comparison of cohorts. Cfr supporting information on statistical plan.

SUMMARY:
This is retrospective research mainly aims to determine the patterns of symptoms, clinical and radiological findings and outcomes in patients with trigeminal neuropathy following trauma or iatrogenic damage and how this translates into costs for the patient and society, work disability and medication use.

The trigeminal nerve and its branches are at risk of damage during multiple dental and maxillofacial procedures: endodontics, extractions, removal of wisdom teeth, implant placement, use of local anaesthesia, orthognatic surgery.

In the event of damage to these nerve branches, there is a high risk of developing a neuropathic pain that is considered very disabling for patients and that interferes with daily activities (eating, drinking, speaking, kissing, etc.). Moreover, there are few medicinal or surgical techniques available to eliminate neuropathy or reduce the symptoms.

Causal procedures (e.g. the removal of wisdom teeth) are among the most frequently performed surgical procedures. The number of injuries increases every year, partly due to an increase in dental procedures. The often relatively minimal intervention combined with the major impact of these injuries on the patient's quality of life sometimes leads to medico-legal actions. The limited symptom control with current therapies of these post-traumatic neuropathies of the trigeminal nerve causes frustration and impotence in both the patient and the attending physician, which can also lead to medical shopping.

Based on chart analysis, this study will examine the causes, possible risk factors and presenting symptoms, how this is reflected in clinical research and examinations, and which treatments are being instituted. Patient records from the Oral and Maxillofacial Surgery department between January 2010 and October 2018 will be checked. In addition, we wish to check the costs incurred by these patients as well as the work disability. To this end, a collaboration is being organised with Christian Mutuality (CM), the largest health insurance provider in Belgium.

In order to increase the power of the study, the clinical data from the already coded, retrospective dataset of Prof. Tara Renton, co-investigator, will be transferred to the dataset of this new study.

ELIGIBILITY:
Inclusion Criteria:

* Presentation with post traumatic, iatrogenic, injury of the trigeminal nerve or its branches (eg. inferior alveolar nerve, lingual nerve)
* Iatrogenic nerve injury caused by M3 removal, implant placement, orthognathic surgery, endodontic therapy, non-M3 removal, local anesthesia injection, trauma.
* Clinical diagnosis of neurosensory deficit in the distribution of the trigeminal nerve caused by a previous dental or maxillofacial procedure in the vicinity of the affected branch.

Exclusion Criteria:

* Neuropathic pain in another region than the trigeminal nerve
* Neuropathic pain not caused by iatrogenic injury

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with post- traumatic, including iatrogenic, injury to branches of the trigeminal nerve seen at the department of Oral & Maxillofacial Surgery at UZ Leuven between January 2010 and October 2018 and possible subsequent post-traumatic neuropathy (PTN). To improve statistical power, the coded dataset from a retrospective study by prof. Tara Renton, co-investigator, will be provided to the principal investigator of the current study (dr. Fréderic Van der Cruyssen) and merged with the dataset acquired in this study to further analyze presentation, symptoms, clinical exam, radiographic evaluation, treatments and outcome parameters. The dataset provided by prof. Tara Renton was build by using the same inclusion and exclusion criteria between January 2010 and October 2018. This should allow for a justified merging of both datasets. Statistical analysis will determine correlation of data.
Sampling Method: Non-Probability Sample
Enrollment: 1333 (Actual)
Dates: Start 2019-01-28 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
Healthcare costs | 10 years
  What is the difference in total healthcare costs per patient and in total in patients with iatrogenic trigeminal nerve injury seen in our department according to cause of injury, injured nerve and outcome (temporary or permanent injury)?
  * A temporary injury will be defined as an injury that completely recovered with no more symptoms and clinical exam parameters within the normal limits during one of the consultations during the follow up period.
  * Permanent injury will be defined as an injury where no significant improvement in symptoms or clinical exam parameters was seen during one of the consultations during the follow up period.
Productivity loss | 10 years
  What is the average productivity loss in days in patients with iatrogenic trigeminal nerve injury seen in our department according to cause of injury, injured nerve and outcome (temporary or permanent injury)?
Medication use | 10 years
  Amount of medication use per medication class per patient in patients with iatrogenic trigeminal nerve injury seen in our department according to cause of injury, injured nerve and outcome (temporary or permanent injury)?

SECONDARY OUTCOMES:
Clinical predictors of persistency | 10 years
  Are symptoms or clinical exam parameters (2 pointdiscrimination, directional sense, light touch, percentage of dermatome affected, pinprick threshold), MRCS classification and Sunderland classification predictive of a temporary or permanent injury? If so, which parameters can be withheld?
Legal action | 10 years
  If data is present in the patient file regarding legal action taken by the patient against the caregiver who caused the injury this will be registered. We will evaluate how many patients undertook legal action and if they received compensation.
Survival analysis | 10 years
  If sufficient follow up data is present, we will evaluate how long symptoms are present in case of a temporary injury and evaluate evolution of symptoms in relation to time.
Influence of imaging on treatment decision | 10 years
  Was imaging performed in light of the injury? If yes, what imaging modality was used (conebeam CT, CT, MRI, orthopantomogram) and did this influence treatment decisions?
PROMS comparison between cohorts | 10 years
  When looking at PROMS questionnaires applied in our department: are the results from the questionnaires comparable between the different causes of nerve injury, different affected branches? Are results comparable between patients suffering from a temporary or permanent injury?
Quality of life between cohorts | 10 years
  Is there a correlation between quality of life measured with EQ5D questionnaire and cause of injury, temporary versus permanent injuries, healthcare costs, productivity loss or medication use?

CONTACTS AND LOCATIONS:
Locations (1):
- dep. Oral & Maxillofacial Surgery, Leuven, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: Undecided
Source data will be directly accessible to the rightful instance or person on request. All medical data, the data collected in the course of the study is treated with the utmost confidentiality. The medical secrecy, the international guidelines (ICH-GCP) and the Belgian legislation are complied with. The investigators undertake to respect the conditions in the European General Data Protection Regulation (Europese Algemene Verordening Gegevensbescherming, AVG) and the Belgian legislation on the protection of natural persons with regard to the processing of personal data.
  The CastorEDC (www.castoredc.com) platform will be used to ensure a systematic approach towards entering datapoints after accessing the patient record. After reading the patient record in KWS, all data will be coded immediately in the CastorEDC database by creating a new and unique identifier, the study ID.

REFERENCES:
- [Background] Klazen Y, Van der Cruyssen F, Vranckx M, Van Vlierberghe M, Politis C, Renton T, Jacobs R. Iatrogenic trigeminal post-traumatic neuropathy: a retrospective two-year cohort study. Int J Oral Maxillofac Surg. 2018 Jun;47(6):789-793. doi: 10.1016/j.ijom.2018.02.004. Epub 2018 Mar 6. PMID 29523381
- [Result] Van der Cruyssen F, Peeters F, Gill T, De Laat A, Jacobs R, Politis C, Renton T. Signs and symptoms, quality of life and psychosocial data in 1331 post-traumatic trigeminal neuropathy patients seen in two tertiary referral centres in two countries. J Oral Rehabil. 2020 Oct;47(10):1212-1221. doi: 10.1111/joor.13058. Epub 2020 Aug 2. PMID 32687637
- [Derived] Van der Cruyssen F, Peeters F, De Laat A, Jacobs R, Politis C, Renton T. Prognostic factors, symptom evolution, and quality of life of posttraumatic trigeminal neuropathy. Pain. 2022 Apr 1;163(4):e557-e571. doi: 10.1097/j.pain.0000000000002408. PMID 34393199
- See also: Study website of the dep. of Oral and Maxillofacial surgery, UZ Leuven, Belgium — http://www.uzleuven.be/nl/mond-kaak-en-aangezichtschirurgie/klinische-studies
- See also: Website of the research group OMFS-IMPATH — https://omfsimpath.be

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-23): https://cdn.clinicaltrials.gov/large-docs/55/NCT04612855/Prot_SAP_000.pdf